CLINICAL TRIAL: NCT06682910
Title: An Early Feasibility Trial to Assess the Safety and Accuracy of the Microtech System in Heart Failure Patients Undergoing Left Ventricular Assist Device Implantation
Brief Title: Assessment of Safety and Accuracy of the Microtech System in Patients Undergoing Left Ventricular Assist Device Implantation
Acronym: Microtech-LVAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Microtech Medical Technologies, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Microtech-001
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Microtech System (Experimental): Microtech System
  Interventions: Device: Microtech sensor pressure

INTERVENTIONS:
Device: Microtech sensor pressure — Microtech sensor implantation

SUMMARY:
The Microtech-LVAD study is designed as a prospective, single arm, multi-center early feasibility study. Approximately 15 patients will be enrolled in the study. The study will be limited to patients in whom it is decided, based on routine clinical practice, that the LVAD will be implanted via a midline sternotomy. In the first 5 study patients, the device will be implanted in the RA; subsequently, the device will be implanted in the LA unless the patient is deemed at high risk of post-LVAD right heart failure, in which case the device will be placed in the RA

DETAILED DESCRIPTION:
The Microtech-LVAD study is designed as a prospective, single arm, multi-center early feasibility study. Approximately 15 patients will be enrolled in the study. The study will be limited to patients in whom it is decided, based on routine clinical practice, that the LVAD will be implanted via a midline sternotomy. In the first 5 study patients, the device will be implanted in the RA; subsequently, the device will be implanted in the LA unless the patient is deemed at high risk of post-LVAD right heart failure, in which case the device will be placed in the RA. Clinical data will be collected pre-operatively, intra-operatively, throughout the post-operative hospitalization period, at discharge and at 1, 3-6, 9 and 12 months post-index procedure

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled to undergo an elective LVAD implantation via midline sternotomy based on routine practice at the participating center.
* Patient is characterized as INTERMACS profile 2 or greater.
* Patient is able and willing to provide written informed consent.
* Patient is willing and able to comply with all required post-procedure follow-up visits.

Exclusion Criteria:

* Pre-operative coagulopathy or thrombocytopenia
* For an intended LA implant, patient has a device implanted in the left atrial appendage (e.g., WATCHMAN or similar device) or a mechanical mitral valve
* Patient has an atrial myxoma
* Patient has pre-operative evidence of thrombus in the chamber in which the device is intended to be implanted
* Patient has a history of stroke or transient ischemic attack within 6 months prior to the index procedure
* History of systemic or pulmonary thromboembolism or deep vein thrombosis (DVT) within the last 6 months
* Patient has a history of congenital heart disease, including known atrial septal defect that is not corrected (including during the LVAD implantation procedure)
* Patient has severe mitral regurgitation (for an LA implant) or severe tricuspid regurgitation (for an RA implant) that is not intended to be corrected during the LVAD implantation
* Patient has known allergy to stainless steel or titanium
* Patient has noncardiac comorbidity that, in the opinion of the Principal Investigator, may limit life expectancy to less than 1 year
* Patient is pregnant or intends to become pregnant prior to completion of all protocol follow-up requirements
* Patient is participating in another investigational study that has not reached its primary endpoint
* Intraoperative identification of any anatomical finding that would preclude safe access to, or closure of, the intended atrial chamber, or fixation of the device within the chamber including, but not limited to:

  1. Identification of thrombus in the atrium in which the device will be implanted
  2. Atrial anatomy deemed to be too thin or fragile to accept the implant
  3. Epicardial adhesions or any intraoperative finding that would complicate access or closure of the atrium in which the device is intended to be implanted

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Co-Primary Efficacy Endpoint | 6 months
  1. Successful deployment of the intracardiac sensor.
  2. Freedom from failure of the Microtech System to obtain valid intracardiac pressures by at least one method (CW/DB), in at least one timepoint up to 6 months.
Co-Primary Safety Endpoint | 1 month
  1. Anatomic stability of the implant assessed by echocardiographic imaging through 1 month.
  2. The incidence of device- or implant procedure-related adverse events through 1 month

SECONDARY OUTCOMES:
The earliest post-operative day at which "valid" pressure measurements can be made from the Microtech implant | 1 month
  The earliest post-operative day at which "valid" pressure measurements can be made from the Microtech implant. A "valid" pressure measurement will be defined as a signal for which the system indicates a "fidelity score" >0.7. Details of the fidelity score are provided in the protocol
Accuracy of Microtech pressure measurements in comparison to those obtained simultaneously by pulmonary artery catheter | pre procedure, 3-6 months
  Accuracy of Microtech pressure measurements in comparison to those obtained simultaneously by pulmonary artery catheter (PAC; LAP from Microtech compared to PCWP from PAC, and RAP from Microtech and RAP from PAC or superior vena caval central line) at baseline and at a follow up between 3- and 6-months post implantation
Accuracy of Microtech pressure measurements in comparison to those obtained simultaneously by pulmonary artery catheter | 1 year
  Accuracy of Microtech pressure measurements in comparison to those obtained simultaneously by pulmonary artery catheter (LAP from Microtech compared to PCWP from PAC, and RAP from Microtech and RAP from PAC or superior vena caval central line) at all follow visits from which data are available throughout the 1 year follow up period
Anatomic stability of the implant over the observation period | post operation, 1 month, 3-6 months, 9 months, 12 months
  Anatomic stability of the implant over the observation period, assessed by echocardiographic imaging at post-op, 1, 3-6, 9, 12 months follow-up visits
The incidence of device-related adverse events | 12 months
  The incidence of device-related adverse events through 1 year follow-up
Correlation of changes of sensor-measured atrial pressure | 1 month, 3-6 months , 9months and 12 month
  Correlation of changes of sensor-measured atrial pressure with the following clinical parameters performed on the 1, 3-6, 9 and 12 month follow up visits:
  1. changes of NTproBNP
  2. changes of KCCQ
  3. episodes of heart failure exacerbations
  4. LVAD suction events
  5. clinical assessments consistent with hypovolemia
  6. changes in pressure measurements during RPM ramp tests
Usability of the system | baseline, 30-6 months, 12 months
  Usability of the system in order to obtain pressure measurements (Human Factors testing) at baseline, 3-6 months and 12 months visits

CONTACTS AND LOCATIONS:
Locations (2):
- Columbia University Medical Center/ NewYork Presbyterian Hospital or CUMC/NYPH, New York, New York, United States
- Rabin Medical Center, Petach Tikvah, Israel

IPD SHARING:
Plan to Share IPD: No